CLINICAL TRIAL: NCT03804242
Title: A Randomized Controlled Trial of a Positive Youth Development Group
Brief Title: Black Youth M.A.T.T.E.R: Positive Youth Development Group Intervention
Acronym: BYM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caitlin Sayegh, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APP-18-07635
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Depression, Anxiety
Keywords: positive youth development; school-to-prison pipeline; mental health stigma; help-seeking; identity
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot trial of intervention versus usual care
Masking Description: Participants, school staff, researchers, and outcome assessor will all be aware of condition assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Youth M.A.T.T.E.R. (Experimental): The session topics are as follows: (1) Debunking the Stigma of Mental Health in the Black Community, (2) School to Prison Pipeline, (3) Achievement Gap, (4) Cultural Barrier that Black Students Experience with Teachers, (5) Trauma 101, (6) Trauma 102, (7) Actions of Today, Blueprints for Tomorrow: Youth Organizing to Transform Education film, (8) My Voice Will Be Heard (Part I), and (9) My Voice Will Be Heard (Part II). The intervention will be conducted in 2-hour weekly group sessions.
  Interventions: Behavioral: Black Youth M.A.T.T.E.R.: Molding Young Advocates While Transforming the School to Prison Pipeline Through Psychological Services Education and Resilience
- Usual Care (No Intervention): All participants already participate in Youth Justice Coalition's Free LA High School. Those in control condition will participate in educational activities as usual.

INTERVENTIONS:
Behavioral: Black Youth M.A.T.T.E.R.: Molding Young Advocates While Transforming the School to Prison Pipeline Through Psychological Services Education and Resilience — This is a group psychoeducational and positive youth development intervention for students who have been expelled from school and are now enrolled in a specialized school at Youth Justice Coalition.
  Arms: Black Youth M.A.T.T.E.R.

SUMMARY:
One in three Black boys born today in the United States will be incarcerated at some point in their lifetime, compared to one in 17 White boys. Black males are more likely to be arrested, convicted, and given unfair sentences. Black youth comprise of 16% of the Nation's public schools, but account for 32% of suspended students. For over 30 years, research has consistently highlighted the disproportionately severe disciplinary practices used with Black male students.Consistent research demonstrates that students who are suspended or expelled tend to drop out of school and/or become incarcerated in a juvenile detention center. Black students may relate their racial-ethnic identity, such as their understanding of their race and ethnicity, to academic success. Moreover, their attitudes may result from the expectation of their teachers. It is imperative that advocates devoted to positive youth development intervene to this issue negatively affecting the well-being of Black youth. Under the mentorship of Caitlin Sayegh, Ph.D., postdoctoral fellow Tierra Ellis, Ph.D., has developed a 9-session group intervention called Black Youth M.A.T.T.E.R. (BYM), which aims to debunk mental health stigma, help children shift their cognitive distortions about education, and normalize their experiences through group activities, while introducing them to advocacy and self-empowerment. This intervention may decrease mental health symptoms, increase motivation to approach goal-oriented outcomes, and reverse internalized beliefs and attitudes which may foster more positive perceptions related to school.

DETAILED DESCRIPTION:
The proposed study is a randomized control trial mixed-methods pilot study of BYM. We aim to finalize the intervention protocol, assess feasibility and acceptability of the intervention, and evaluate the potential impact of BYM on pilot participants. The mixed-methods research design approach will be used within a single study for the collection, analyzing, and merging of qualitative and quantitative data. The purpose of a convergent parallel mixed methods research design is to simultaneously collect qualitative and quantitative data for a more comprehensive analysis.

Research Questions: (1) What do Black adolescents and other community stakeholders perceive as the most effective approaches for the BYM project? (2) What are BYM participants' perceptions of the intervention? (3) Is there a decrease in mental health symptoms (e.g., depression, anxiety, trauma) for BYM participants? (3) Is there an increase in resiliency for BYM participants? (4) Is there an increase in positive attitudes toward seeking mental health treatment for BYM participants? (5) Is there a difference in motivation to approach goal-oriented outcomes for BYM participants? (6) Is there an increase in perceived positive self-concept for BYM participants? (7) Is there a decrease in risk behaviors for BYM participants? Intervention Description: The session topics are as follows: (1) Debunking the Stigma of Mental Health in the Black Community, (2) School to Prison Pipeline, (3) Achievement Gap, (4) Cultural Barrier that Black Students Experience with Teachers, (5) Trauma 101, (6) Trauma 102, (7) Actions of Today, Blueprints for Tomorrow: Youth Organizing to Transform Education film, (8) My Voice Will Be Heard (Part I), and (9) My Voice Will Be Heard (Part II). The intervention will be conducted in 2-hour weekly group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Black adolescents attending Youth Justice Coalition Free LA High School who have been suspended or expelled from their respective schools due to behavioral problems

Exclusion Criteria:

* Active psychosis or suicidal ideation

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms and anxiety symptoms | 61 weeks
  Revised Children's Anxiety and Depression Scale. The T-score related to Total Anxiety and Depression score will be examined (ranging from 26 to >80). Higher scores indicate increased depression and anxiety symptoms.
Change in trauma symptoms | 61 weeks
  Trauma Symptom Checklist for Children: Examining Posttraumatic Stress T-score (ranging from 26 to >80), where higher scores indicated greater PTSD symptoms.
Change in Youth Reporting Substance Use | 61 weeks
  Youth Risk Behavior Survey. We will examine dichotomous use of tobacco, alcohol, cannabis, and other drugs

SECONDARY OUTCOMES:
Change in Resiliency | 61 weeks
  Resiliency Scale; range from 0 to 14 with higher scores representing more resiliency
Change in Levels of Help-Seeking | 61 weeks
  Attitudes Toward Seeking Professional Help; scores range from 0 to 30 with higher scores indicated more positive views of help-seeking

IPD SHARING:
Plan to Share IPD: No